CLINICAL TRIAL: NCT06205407
Title: A Single-dose, Open-label, Randomized, 2-way, Cross-over Pivotal Bioequivalence Study to Qualify Manufacturing Site Transfer From Viatris to Neolpharma, for Spironolactone/Hydrochlorothiazide Film Coated Tablets in Healthy Adult Participants Under Fasted Conditions.
Brief Title: A Study to Learn How the Body Processes Spironolactone and Hydrochlorothiazide Film Coated Tablets Manufactured at Two Sites: Viatris and Neolpharma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B9531002; NCT06205407 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-01-02; First posted 2024-01-16 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants
Keywords: Phase I; Pharmacokinetics; Spironolactone/Hydrochlorothiazide film coated tablets; Bioequivalence
MeSH Terms: interventions — Spironolactone; Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: This will be an open-label, randomized, single-dose, 2-treatment, 2-period, 2-sequence, crossover study in adult healthy male and/or female participants. Approximately 40 participants will be enrolled in the study (20 in each treatment sequence).
  There will be a minimum 4-day washout period between successive doses (ie, administration of subsequent doses of study medication will not occur until at least 4 days after the previous dose of study medication).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A (Active Comparator): Spironolactone/Hydrochlorothiazide (25 mg/25 mg) film coated tablets manufactured at Viatris.
  Interventions: Drug: Spironolactone/Hydrochlorothiazide (25 mg/25 mg) film coated tablets from Viatris
- Treatment B (Experimental): Spironolactone/Hydrochlorothiazide (25 mg/25 mg) film coated tablets manufactured at Neolpharma.
  Interventions: Drug: Spironolactone/Hydrochlorothiazide (25 mg/25 mg) film coated tablets from Neolpharma.

INTERVENTIONS:
Drug: Spironolactone/Hydrochlorothiazide (25 mg/25 mg) film coated tablets from Viatris — Manufactured at Viatris
  Arms: Treatment A
Drug: Spironolactone/Hydrochlorothiazide (25 mg/25 mg) film coated tablets from Neolpharma. — Manufactured at Neolpharma.
  Arms: Treatment B

SUMMARY:
The purpose of the study is to understand how the body processes Spironolactone and Hydrochlorothiazide after taking Spironolactone and Hydrochlorothiazide film coated tablets manufactured at two sites: Viatris and Neolpharma by mouth.

The study is seeking for:

* Both male and female participants.
* participants who must be 18 to 75 years of age.
* Body Mass Index of participants should be 16 to 32 kilogram per meter squared and body weight should be more than 50 kilograms (110 pounds).

About 40 participants will enter the study (20 in each group). Study consists of two periods. On Day 1 of each period, participants will receive a single amount of Spironolactone and Hydrochlorothiazide tablets. The total duration of study will be 71 days. Follow up may occur via telephone after 35 days after taking the final tablet of the study medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 75 years of age, inclusive, at the time of signing the ICD.
2. BMI of 16-32 kg/m2; and a total body weight >50 kg (110 lb).
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

   1. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
   2. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
2. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
4. Current use of any prohibited concomitant medication(s) or participant unwilling or unable to use a required concomitant medication(s).
5. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
6. A positive urine drug test. A single repeat for positive drug screen may be allowed.
7. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If systolic BP is ≥ 140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
8. Hepatic dysfunction defined as:

   1. Total bilirubin ≥1.5 × ULN (For Gilbert's syndrome, direct bilirubin >ULN is exclusionary)
   2. AST ≥1.5 × ULN
   3. ALT ≥1.5 × ULN
9. Baseline standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms). If QTcF exceeds 450 ms, the ECG should be repeated twice and the average of the 3 QTcF values used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
10. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
11. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
12. History of sensitivity to heparin or heparin induced thrombocytopenia.
13. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
14. History of hypersensitivity to spironolactone or HCTZ or any of the components in the formulation of the study products, or allergic to thiazide diuretics or to other sulfonamide-derived drugs.
15. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Clinical Trials of Texas, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9531002

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Treatment A Followed by Treatment B: Participants randomized to sequence 1 received spironolactone/hydrochlorothiazide 25/25 milligram (mg) film coated tablets manufactured at Viatris (Treatment A) and Neolpharma (Treatment B) on Day 1 of Period 1 and Period 2, respectively. A washout period of at least 4 days was maintained between each treatment period.
- Sequence 2: Treatment B Followed by Treatment A: Participants randomized to sequence 2 received spironolactone/hydrochlorothiazide 25/25 mg film coated tablets manufactured at Neolpharma (Treatment B) and Viatris (Treatment A) on Day 1 of Period 1 and Period 2, respectively. A washout period of at least 4 days was maintained between each treatment period.
Period: Period 1
Arm/Group | Sequence 1: Treatment A Followed by Treatment B | Sequence 2: Treatment B Followed by Treatment A
Started | 21 | 21
Treated | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Washout
Arm/Group | Sequence 1: Treatment A Followed by Treatment B | Sequence 2: Treatment B Followed by Treatment A
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence 1: Treatment A Followed by Treatment B | Sequence 2: Treatment B Followed by Treatment A
Started | 21 | 21
Treated | 19 | 20
Completed | 19 | 19
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study intervention.
Groups:
- All Participants: Participants randomized to sequence 1 received spironolactone/hydrochlorothiazide 25/25 mg film coated tablets manufactured at Viatris and Neolpharma in Period 1 and 2, respectively. Participants randomized to sequence 2 received Spironolactone/Hydrochlorothiazide 25/25 mg film coated tablets manufactured at Neolpharma and Viatris in Period 1 and 2, respectively. A washout period of at least 4 days was maintained between each treatment period.
Arm/Group | All Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.4 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30
  Black or African American | 11
  American Indian or Alaska Native | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Spironolactone and Hydrochlorothiazide Following a Single Oral Dose of Spironolactone/Hydrochlorothiazide 25/25 mg Film Coated Tablet Manufactured at Viatris
Description: Maximum plasma concentration of Spironolactone and Hydrochlorothiazide after participants received a single oral dose of 25/25 mg film coated tablets manufactured at Viatris.
Time Frame: Pre-dose (0 hours [hrs]) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hrs post dose
Population: All participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Treatment A: Participants randomized to sequences 1 and 2 received spironolactone/hydrochlorothiazide 25/25 mg film coated tablets manufactured at Viatris in Period 1 and 2, respectively.
Arm/Group | Treatment A
Number analyzed (Participants) | 41
nanogram per milliliter (ng/mL)
  Spironolactone | 28.73 (52)
  Hydrochlorothiazide | 177.8 (33)

2. Primary Outcome: Cmax of Spironolactone and Hydrochlorothiazide Following a Single Oral Dose of Spironolactone/Hydrochlorothiazide 25/25 mg Film Coated Tablet Manufactured at Neolpharma
Description: Maximum plasma concentration of Spironolactone and Hydrochlorothiazide after participants received a single oral dose of 25/25 mg film coated tablets manufactured at Neolpharma.
Time Frame: Pre-dose (0 hrs) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hrs post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Treatment B: Participants randomized to sequences 1 and 2 received spironolactone/hydrochlorothiazide 25/25 mg film coated tablets manufactured at Neolpharma in Period 1 and 2, respectively.
Arm/Group | Treatment B
Number analyzed (Participants) | 40
nanogram per milliliter (ng/mL)
  Spironolactone | 25.57 (47)
  Hydrochlorothiazide | 179.2 (33)

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUCinf) of Spironolactone and Hydrochlorothiazide Following a Single Oral Dose of Spironolactone/Hydrochlorothiazide 25/25 mg Film Coated Tablet Manufactured at Viatris
Description: AUCinf was defined as area under the plasma concentration-time profile from time 0 extrapolated to infinite time. Area under the plasma concentration-time curve from time zero to infinity of Spironolactone and Hydrochlorothiazide after participants received a single oral dose of 25/25 mg film coated tablets manufactured at Viatris.
Time Frame: Pre-dose (0 hrs) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hrs post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Treatment A
Number analyzed (Participants) | 41
nanogram*hour per milliliter (ng*hr/mL)
  Spironolactone | 53.60 (44)
  Hydrochlorothiazide | 1269 (27)

4. Primary Outcome: AUCinf of Spironolactone and Hydrochlorothiazide Following a Single Oral Dose of Spironolactone/Hydrochlorothiazide 25/25 mg Film Coated Tablet Manufactured at Neolpharma
Description: AUCinf was defined as area under the plasma concentration-time profile from time 0 extrapolated to infinite time. Area under the plasma concentration-time curve from time zero to infinity of Spironolactone and Hydrochlorothiazide after participants received a single oral dose of 25/25 mg film coated tablets manufactured at Neolpharma.
Time Frame: Pre-dose (0 hrs) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hrs post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment B
Number analyzed (Participants) | 40
ng*hr/mL
  Spironolactone | 52.52 (40)
  Hydrochlorothiazide | 1281 (32)

5. Secondary Outcome: Plasma Elimination Half Life (t1/2) of Spironolactone and Hydrochlorothiazide Following a Single Oral Dose of Spironolactone/Hydrochlorothiazide 25/25 mg Film Coated Tablet Manufactured at Viatris
Description: t1/2 was defined as terminal elimination half-life. Plasma elimination half life of Spironolactone and Hydrochlorothiazide after participants received a single oral dose of 25/25 mg film coated tablets manufactured at Viatris.
Time Frame: Pre-dose (hrs) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hrs post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Treatment A
Number analyzed (Participants) | 41
Hour
  Spironolactone | 2.252 (1.3694)
  Hydrochlorothiazide | 10.91 (2.1620)

6. Secondary Outcome: t1/2 of Spironolactone and Hydrochlorothiazide Following a Single Oral Dose of Spironolactone/Hydrochlorothiazide 25/25 mg Film Coated Tablet Manufactured at Neolpharma
Description: t1/2 was defined as terminal elimination half-life. Plasma elimination half-life of Spironolactone and Hydrochlorothiazide after participants received a single oral dose of 25/25 mg film coated tablets manufactured at Neolpharma.
Time Frame: Pre-dose (0 hrs) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hrs post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Treatment B
Number analyzed (Participants) | 40
Hour
  Spironolactone | 2.413 (1.9284)
  Hydrochlorothiazide | 10.17 (1.7661)

7. Secondary Outcome: Time to Reach Cmax (Tmax) of Spironolactone and Hydrochlorothiazide Following a Single Oral Dose of Spironolactone/Hydrochlorothiazide 25/25 mg Film Coated Tablet Manufactured at Viatris
Description: Time to reach maximum concentration of Spironolactone and Hydrochlorothiazide after participants received a single oral dose of 25/25 mg film coated tablets manufactured at Viatris.
Time Frame: Pre-dose (0 hrs) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hrs post dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A
Number analyzed (Participants) | 41
Hour
  Spironolactone | 1.00 [0.500 to 3.00]
  Hydrochlorothiazide | 2.48 [1.00 to 4.00]

8. Secondary Outcome: Tmax of Spironolactone and Hydrochlorothiazide Following a Single Oral Dose of Spironolactone/Hydrochlorothiazide 25/25 mg Film Coated Tablet Manufactured at Neolpharma
Description: Time to reach maximum concentration of Spironolactone and Hydrochlorothiazide after participants received a single oral dose of 25/25 mg film coated tablets manufactured at Neolpharma.
Time Frame: Pre-dose (0 hrs) and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hrs post dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment B
Number analyzed (Participants) | 40
Hour
  Spironolactone | 1.00 [0.417 to 3.97]
  Hydrochlorothiazide | 2.00 [1.02 to 4.05]

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Any adverse events occurring following start of treatment were considered as treatment emergent adverse event (TEAE). Treatment-related TEAEs were determined by the investigator. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect.
Time Frame: From Baseline up to 35 days after the last dose of study intervention (approximately 41 days)
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment A: Participants randomized to sequences 1 and 2 received spironolactone/hydrochlorothiazide 25/25 mg film coated tablets manufactured at Viatris in Period 1 and 2, respectively. A washout period of at least 4 days was maintained between each treatment period.
- Treatment B: Participants randomized to sequences 1 and 2 received spironolactone/hydrochlorothiazide 25/25 mg film coated tablets manufactured at Neolpharma in Period 1 and 2, respectively. A washout period of at least 4 days was maintained between each treatment period.
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 41 | 40
Participants
  All-causality TEAE | 8 | 8
  Treatment-related TEAE | 5 | 2
  All-causality SAE | 0 | 0

10. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities Meeting AE Criteria (Without Regard to Baseline Abnormality)
Description: Abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) that met AE reporting criteria were those that worsened from baseline and considered clinically significant in the medical and scientific judgment of the investigator. Laboratory abnormalities that met any of the following conditions must be reported as an AE: (1) was associated with accompanying symptoms; (2) required additional diagnostic testing or medical/surgical intervention; (3) led to a change in study dosing (outside of any protocol-specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy.
Time Frame: From Baseline up to 35 days after the last dose of study intervention (approximately 41 days)
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 41 | 40
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Vital Signs Data Meeting AE Criteria
Description: Abnormal vital sign measurement results (supine blood pressure, pulse rate) that met AE reporting criteria were those that worsened from baseline and considered clinically significant in the medical and scientific judgment of the investigator. Vital sign abnormalities that met any of the following conditions must be reported as an AE: (1) was associated with accompanying symptoms; (2) required additional diagnostic testing or medical/surgical intervention; (3) led to a change in study dosing (outside of any protocol-specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy.
Time Frame: From Baseline up to 35 days after the last dose of study intervention (approximately 41 days)
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 41 | 40
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting AE Criteria
Description: Abnormal ECG results meeting AE reporting criteria were those that worsened from baseline, and considered clinically significant in the medical and scientific judgment of the investigator. ECG findings that may qualify as AE included: marked sinus bradycardia (rate <40 beats per minute [bpm]) lasting minutes; new PR interval prolongation >280 millisecond (ms); new prolongation of QT interval corrected using Fridericia's formula (QTcF) to >480 ms (absolute); new prolongation of QTcF by >60 ms from baseline; new onset atrial flutter or fibrillation, with controlled ventricular response rate: i.e., rate <120 bpm; new onset type I second degree (Wenckebach) atrioventricular (AV) block of >30-second duration; frequent premature ventricular contraction/complex (PVC), triplets, or short intervals (<30 seconds) of consecutive ventricular complexes.
Time Frame: From Baseline up to 35 days after the last dose of study intervention (approximately 41 days)
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 41 | 40
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to 35 days after the last dose of study intervention (approximately 41 days)
Description: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Arm/Group | Treatment A | Treatment B
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 8/41 | 8/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=41) | Treatment B (N=40)
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 4 | 5
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT06205407/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT06205407/SAP_001.pdf